CLINICAL TRIAL: NCT02128581
Title: A Dose-response Study of the Effects of Exendin-9,39 on Gastrointestinal Symptoms and Food Intake.
Brief Title: A Dose-response of the Effects of Exendin-9,39 on GI Symptoms and Food Intake
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Adrian Vella, Consultant, Endocrinology, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14-002150; R01DK082396 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2014-04-18; First posted 2014-05-01 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Diabetes; Roux-en-Y Gastric Bypass
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saline (Placebo Comparator): a saline infusion will be started and maintained till the end of the study at 1300 (300 minutes).
  Interventions: Other: Saline
- Exendin-9,39 @ 300 (Active Comparator): Exendin-9,39 @ 300pmol/kg/min
  Interventions: Drug: Exendin-9,39
- Exendin-9,39 @ 750 (Active Comparator): Exendin-9,39 @ 750pmol/kg/min
  Interventions: Drug: Exendin-9,39

INTERVENTIONS:
Drug: Exendin-9,39 — use Exendin-9,39 @ 750pmol/kg/min and Exendin-9,39 @ 300pmol/kg/min to block endogenous GLP-1 in humans after gastric bypass and determine contribution of GLP to satiety after meal ingestion
  Arms: Exendin-9,39 @ 300; Exendin-9,39 @ 750
Other: Saline
  Arms: Saline

SUMMARY:
Exendin-(9,39) has been shown to have effects on beta-cell function, and after gastric bypass, to accelerate gastrointestinal transit. - infused at rates of 300pmol/kg/min. Given that gastrointestinal transit is typically delayed by Glucagon-Like Peptide-1 (GLP-1) and also that this hormone causes decreased food intake through increased satiation, it is reasonable to expect an effect of Exendin-9,39 on appetite. This may help explain the effects of gastric bypass on food intake. To examine the effect of Exendin on food intake we propose a dose-response study to determine whether the compound has effects in a dose-dependent fashion. We will examine the presence of gastrointestinal symptoms as well as food intake in the immediate aftermath of a test meal and the subsequent hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have undergone Roux en-Y Gastric Bypass at least 6 months prior to enrollment in the study.
* Subjects without active systemic illness.

Exclusion Criteria:

* Subjects <20 years of age will not be studied to minimize the possibility of type 1 diabetes.
* Subjects >70 years of age will not be studied to minimize the potential confounding effects of age on glucose tolerance.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Calories consumed during buffet meal test | approximately 300 minutes after initiation
  The calories consumed during buffet meal test at the end of each study test will help determine the effect of GLP-1 receptor blockade with Exendin-9,39 on food intake.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials